CLINICAL TRIAL: NCT06402851
Title: A Randomized Clinical Trial Comparing Three Anti-Thrombotic Strategies for Patients with Atrial Fibrillation and Severe Chronic Kidney Dysfunction
Brief Title: Vitamin K AntagonISt, Factor Xa Inhibitor or No Anticoagulation in Atrial Fibrillation and DIalytic End-stage Renal DiseasE (VISIONAIRE)
Acronym: VISIONAIRE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVAP-NG 3353
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Atrium; Fibrillation; Chronic Kidney Diseases
Keywords: atrial fibrillation; atrial flutter; oral anticoagulation; dialysis
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency, Chronic; Atrial Flutter | interventions — Anticoagulants; edoxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in 1:1:2 to warfarin, edoxaban or no OAC, stratified by renal replacement status.
Who Masked: Outcomes Assessor
Masking Description: All study endpoints will be assessed by an independent Clinical Events Committee (CEC), whose members will be unaware of randomized treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Warfarin (Active Comparator): Full-dose anticoagulation with adjusted dose (target INR 2.0-3.0) warfarin.
  Interventions: Drug: Anticoagulant Oral
- Edoxaban (Experimental): Dose will be based on label from Brazil considering adjustment for low CrCl, that is, 30 mg QD.
  Interventions: Drug: Anticoagulant Oral
- No anticoagulation (No Intervention): No oral anticoagulation should be used

INTERVENTIONS:
Drug: Anticoagulant Oral — Patients will be anticoagulated following with 30 mg QD edoxaban or adjusted dose warfarin for a target INR 2.0-3.0.
  Other Names: Edoxaban; Warfarin
  Arms: Edoxaban; Warfarin

SUMMARY:
VISIONAIRE (Vitamin K AntagonISt, Factor Xa Inhibitor Or Nothing In Atrial Fibrillation And DIalytic End-stage Renal DiseasE) trial will be a prospective randomized open-label with blinded endpoint adjudication trial including 1500 patients with atrial fibrillation or atrial flutter and advanced chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical atrial fibrillation or flutter (persistent, paroxysmal or permanent);
* CHA2DS2-Vasc ≥ 2 points (≥ 3 if female);
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) ≤ 15 ml/min/1.73 m2 by the CKD-EPI equation (confirmed by two lab results at least 3 months apart) or on chronic renal replacement therapy (Of note: number of patients included in no renal replacement therapy stratum will be capped at around 30% from the total study population).

Exclusion Criteria:

* Active bleeding or severe bleeding < 1 month;
* Prior kidney transplantation;
* Refusal de provide consent
* Severe chronic liver disease (Child C);
* Other indication of oral anticoagulation (e.g.,: venous thromboembolism or pulmonary embolism);
* Prior intracranial hemorrhage;
* Bleeding disorder (other than uremia);
* Platelet count < 50,000 / mm3 ;
* Pregnancy or breastfeeding;
* Mechanical valvar prosthesis;
* Moderate to severe mitral stenosis;
* Need for antithrombotic drugs other than single antiplatelet agents, or need for dual antiplatelet therapy with aspirin plus an ADP receptor blocker;
* Any comorbidity beyond CKD and CV disease (e.g., metastatic cancer) which, in the investigator´s opinion, may impact survival in 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 24 months (median follow-up)
  Time to first occurrence of the composite of stroke or systemic embolism
Primary safety endpoint: | 24 months (median follow-up)
  Major or clinically relevant non-major bleeding according to the ISTH criteria

SECONDARY OUTCOMES:
Secondary efficacy endpoints | 24 months (median follow-up)
  Time to first occurrence of the composite of: death, ischemic or undetermined stroke, or systemic embolism
Secondary efficacy endpoints | 24 months (median follow-up)
  Time to first occurrence of the composite of: CV death, MI, or stroke
Secondary efficacy endpoints | 24 months (median follow-up)
  Time to first occurrence of the composite of: all-cause death, MI, systemic embolism, or stroke
Secondary efficacy endpoints | 24 months (median follow-up)
  All cause death
Secondary safety endpoint | 24 months (median follow-up)
  Time to first occurrence of major bleeding (ISTH)
Secondary safety endpoint | 24 months (median follow-up)
  Time to first occurrence of GUSTO moderate or severe bleeding
Secondary safety endpoint | 24 months (median follow-up)
  Time to first occurrence of TIMI minor and major bleeding
Secondary safety endpoint | 24 months (median follow-up)
  Fatal or intra-cranial bleeding
Net clinical endpoint | 24 months (median follow-up)
  Time to first occurrence of CV death, MI, stroke, systemic embolism, fatal bleeding or bleeding into a critical organ

OTHER OUTCOMES:
Exploratory endpoint | 12 months
  Quality of life by EQ-5D
Exploratory endpoint | 24 months (median follow-up)
  Access site bleeding
Exploratory endpoint | 24 months (median follow-up)
  Fistula or catheter thrombosis
Exploratory endpoint | 24 months (median follow-up)
  Fistula or catheter failure

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto de Cardiologia do DF, Brasília, Federal District
  - Hospital Universitário Maria Aparecida Pedrossian - EBSERH, Campo Grande, Mato Grosso do Sul
  - Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista
  - Santa Casa de Misericórdia de Ponta Grossa, Ponta Grossa

IPD SHARING:
Plan to Share IPD: No
After publication of study primary results in a peer-reviewed scientific medical journal, interested parts in data sharing are welcome to contact the corresponding author directly.